CLINICAL TRIAL: NCT00955097
Title: Evaluation of Intra-operative Ultrasound Contrast Enhancement in the Evaluation of Liver Tumors
Acronym: Definity®
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding for this study
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Robert C. Martin, MD, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Definity 08.0119; 08.0119
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Liver Tumors
Keywords: Definity; liver tumors; intra operative contrast; liver cancer; hepatic tumors; identify liver tumors; surgery liver tumors; Patients with known hepatic tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Definity Contrast Dye (Experimental): During liver surgery Definity contrast dye will be administered follwed by an ultrasound to better detect liver tumors
  Interventions: Drug: Definity®

INTERVENTIONS:
Drug: Definity® — Definity® injections given both pre-ablation and post-ablation

SUMMARY:
The primary purpose of this study is to demonstrate the safety and effectiveness of using an intra-operative ultrasound contrast agent(Definity®) for the identification of known liver tumors.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the safety of the use of intra-operative ultrasound contrast (Definity®) administration. The secondary objective of this study is to demonstrate the improved image quality and conspicuity of known liver tumors using contrast enhancement.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing a hepatic resection or hepatic ablation of pre-operative visualized liver tumor:
2. ≥ 18 years of age
3. If female of child-bearing potential, negative pregnancy test within 14 days prior to surgery
4. If subject is a sexually active male or a sexually active female of child-bearing potential, subject agrees to use a medically accepted form of contraception from the time of enrollment to completion of all follow-up study visits.
5. IRB-approved informed consent, signed by the subject or the subject's legally authorized representative. ≥ 18 years of age

Exclusion Criteria:

1. Not a suitable candidate for operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
adverse events | 6-weeks post surgery
identification of liver tumors | intra-operative

SECONDARY OUTCOMES:
improved ablation of liver tumors | 6-weeks post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martin, MD, Principal Investigator — University of Louisville
Locations (2):
- United States (2):
  - Norton Healthcare, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky